CLINICAL TRIAL: NCT00255359
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled, Dose Escalation Study of the Safety and Efficacy of XTL 2125 in Adult HCV-Infected Patients With Compensated Liver Disease, Who Are Interferon-Alpha Non-Responders or Have Relapsed From Interferon-Alpha Therapy
Brief Title: Safety, Tolerability and Efficacy of XTL 2125 in HCV-Infected Patients Who Are Interferon-Alpha Non-Responders or Relapsers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: XTL Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200517-HMO-CTIL
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Hepatitis C Virus Infection

INTERVENTIONS:
Drug: XTL-2125

SUMMARY:
The study will be a randomized, double blind, placebo controlled, dose rising study in Interferon alpha (IFN-alpha) non-responder HCV infected patients or HCV patients who have relapsed following IFN-alpha therapy. Eligible subjects must have compensated liver disease and serum HCV RNA concentrations above 100,000 IU/mL at screening. The study will include both a single dose period for the evaluation of acute toxicity and single dose pharmacokinetics and a consecutive multi-dose period for the determination of longer-term safety, multiple-dose pharmacokinetics and antiviral activity. The objectives of this study are to evaluate the safety, tolerability, and antiviral activity of escalating single and multiple doses of XTL 2125 in patients with chronic hepatitis C virus infection and to assess the single- and multiple-dose pharmacokinetics of XTL 2125

DETAILED DESCRIPTION:
The study will be of a randomized, double blind, placebo controlled, multicenter design with sequential ascending doses of XTL 2125 in HCV-infected patients with compensated liver disease who did not respond to IFN-alpha therapy or relapsed following this therapy.

This study will include both a single dose session and a multiple dose session. In the single dose session, patients will be randomized to receive a single oral dose of either XTL 2125 or placebo on Day 1, in a dose-escalating design, followed by a multiple dose session that will start on day 8 and will continue for 14 days. The same patients will receive XTL 2125 three times daily at the same dose administered in the single dose session.

The following doses will be administered to groups of 8 patients each: 10 mg, 25 mg, 50 mg, 150 mg, 300 mg and 450 mg. Within each group, 6 subjects will receive XTL 2125 and 2 subjects will receive placebo. No patient will be enrolled in more than one dose level. Doses should be administered one hour before meals with 240 cc water.

Additional patients may be enrolled at previous or intermediate doses to obtain additional safety or pharmacokinetic/pharmacodynamic data and to more accurately define the Maximum Tolerated Dose (MTD).

The MTD will be defined as the last dose level that is successfully administered with a decision to escalate to the next level. If the decision not to escalate to the next level is made then a cohort that receives XTL 2125 at a dose half-way between the last tolerated dose and the non-tolerated dose may be enrolled at the discretion of the Sponsor. If this dose is successfully administered without violating the dose escalation rules, then this interim dose will be considered the MTD.

Six dose cohorts will be prospectively indicated, although additional cohorts may be scheduled at intermediate doses if warranted by the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand and be willing to give written informed consent prior to any study procedures or evaluations and be willing to adhere to all study schedules and requirements.
* Adults 18 to 70 years of age.
* Documented history of positive HCV serology.
* Compensated liver disease as defined by the following at screening: PT greater or equal to 60%, INR < 1.5, serum albumin greater or equal 3.4 g%, and serum bilirubin < 2 mg% (unless dx of Gilbert's Syndrome).
* Serum HCV RNA greater or equal 100,000 IU/mL at screening.
* Patients who were treated and did not respond to IFN-alpha therapy or who withdrew from this therapy within 30 days prior to screening.
* Patients who had completed a fully prescribed course of an approved IFN alpha -based treatment and relapsed following the end of the treatment.
* Patients must be sterile or infertile or use an approved method of contraception from the time that the first dose of study medication is taken until three months following study completion or discontinuation.
* Screening labs as follows: platelet count greater or equal 120,000/mm3; ANC greater or equal 1000/mm3; hemoglobin greater or equal 11.0 g/dL for females and greater or equal 12.0 g/dL for males; serum ALT within normal limits or < 5 x ULN.
* Alpha fetoprotein <25 microg/L at screening.

Exclusion Criteria:

* Any history of significant cardiac, renal, neurologic, metabolic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease other than hepatitis C or any other disease which in the judgment of the investigator would interfere with the study or confound the results.
* Patients with positive HIV serology or positive HBsAg at screening.
* Patients who were not treated previously with the current approved therapy against HCV.
* Patients who have received any previous treatment for HCV infection other than an approved regimen of IFN alpha and ribavirin within 30 days prior to screening.
* Patients with decompensated liver disease or evidence of advanced liver disease such as the presence of ascites, bleeding varices or hepatic encephalopathy.
* Female patients who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* History of alcohol or drug abuse within 6 months of screening.
* Patients who have a positive urine drug screen for substances of abuse (benzodiazepine, THC, opiates, amphetamines, cocaine) at the screening.
* Patients with poor venous access
* History or evidence of hepatocellular carcinoma (HCC).
* Use of prescription or non-prescription drugs that are known to be metabolized in the liver and can potentially interfere with the study medication (such as Marcolide antibiotics, azole antifungals, warfarin, carbamazepine, cyclosporine, midazolam, phenytoin, valporic acid, chlorpromazine, rifampin, quinidine, diazepam and digoxin) 90 days prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Study Completion 2007-11

PRIMARY OUTCOMES:
Safety:
• adverse events, serious adverse events
• laboratory abnormalities by highest toxicity grade
• laboratory abnormalities by largest increase in toxicity grade from baseline
Efficacy:
• Median change from baseline in serum HCV RNA (log10 IU/mL) at day 22.
• Median maximum change from baseline at any time between Day 8 and Day 22.
• Median change from baseline in serum ALT at day 22.
• Percent of patients within each cohort with serum HCV RNA declining at least a 1 log10 from baseline at any assessment between Day 8 and 22.
• AUC using the trapezoidal rule, minus baseline for serum HCV RNA (in the log10 scale) through day 22 (defined as DAVG22).
• Median rate of decline in serum HCV RNA (log10 IU/mL/day) through day 22.
• Median rate of change in serum HCV RNA (log10 IU/mL/day) from day 22 (after the last administration) through day 50 (rebound).
• Median change from day 22 (after the last administration) in serum HCV RNA (log10 IU/mL) at day 50 (rebound).
• Descriptive analysis of changes in the HCV genome (NS5B region coding for RNA dependent RNA polymerase) that may be associated with two weeks of
XTL 2125 monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Eithan Galun, MD, Principal Investigator — Hadassah Medical Organization; Shlomo Dagan, PhD, Study Director — XTL Biopharmaceuticals
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel